CLINICAL TRIAL: NCT07009704
Title: Real-time Continuous Glucose Monitoring and Mobile-based Social Support to Promote Glucose Management During Pregnancy
Brief Title: Glucose Empowerment Through Monitoring and Social Support in Pregnancy
Acronym: GEMS-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005143; K12HD092535 (NIH); K12AR084217 (NIH)
Record Dates: First submitted 2025-01-07; First posted 2025-06-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy, Complications; Gestational Diabetes
Keywords: pregnancy; gestational diabetes; GDM; intervention; hyperglycemia; group chat; continuous glucose monitoring; mobile-based; behavioral change; CGM
MeSH Terms: conditions — Pregnancy Complications; Diabetes, Gestational; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups. Group 1 will receive real-time continuous glucose monitoring plus mobile-based social support. Group 2 will only receive real-time continuous glucose monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Group chat intervention (Experimental): Participants in group 1 will be randomized to wear a real-time continuous glucose monitor for 14 days and participate in a secure mobile-based group chat where they will provide and receive social support for glucose management. Participants will be in the group chat for 60 days.
  Interventions: Behavioral: Mobile-based social support; Behavioral: Real-time continuous glucose monitoring
- Group 2- No group chat intervention (Experimental): Participants in group 2 will be randomized to wear a real-time continuous glucose monitor for 14 days.
  Interventions: Behavioral: Real-time continuous glucose monitoring

INTERVENTIONS:
Behavioral: Mobile-based social support — Participants will be invited to join an encrypted group chat where they will be encouraged to provide and receive social support related to glucose management during early pregnancy. Other study participants and study team members will be in the group chat.
  Arms: Group 1- Group chat intervention
Behavioral: Real-time continuous glucose monitoring — Participants will receive a real-time continuous glucose monitor that pairs with an existing smartphone app that shows minute-by-minute glucose levels and records glucose levels in 5 minute increments.

SUMMARY:
The purpose of the research is to learn whether wearing a continuous glucose monitor that shows blood glucose levels in real time on a smart phone app and participating in a group chat with other research participants will help participants keep a healthy blood glucose level during pregnancy.

High levels of blood glucose during pregnancy can lead to health problems during and after pregnancy. It may also increase the risk for health problems for the developing baby.

The investigators think our program might be a new way to help some people maintain a healthy blood glucose level during pregnancy. When pregnant people know their blood glucose levels are high, they can do things like exercise or drink water to bring their blood glucose levels down. They can also learn what foods to eat to maintain healthy blood glucose levels, and what foods to avoid. The investigators think being in a group chat with other pregnant individuals will allow participants to support and learn from each other. Pregnant individuals should also work with their healthcare providers to manage their blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (<20w0d)
* At least 18 years to 45 years old
* BMI >25, personal history of GDM, or first-degree family member with type II diabetes
* Comfortable conversing in English
* Own a smartphone and willing to use the CGM app and Signal
* Receiving prenatal care and planning to deliver at Tufts Medicine (Boston)
* Signed the consent form
* Currently located in the United States

Exclusion Criteria:

* Current pregnancy a multiple gestation (e.g., twins)
* Smoked during this current pregnancy
* Active hepatitis or HIV infection
* Current pregnancy have any documented fetal congenital anomalies
* Current history of heroin, cocaine, crack, LSD, or methamphetamines
* Current history of alcohol abuse
* Previous gastric bypass
* Shift work that alters the sleep/wake periods
* Have known rheumatological or chronic inflammatory state (i.e., arthritis, inflammatory bowel disease)?
* Chronic illnesses, including diabetes and dialysis, that require regular medication use
* Uncontrolled hypothyroidism
* Known culture of positive chorioamnionitis?
* An adult who is unable to consent (e.g., cognitively impaired adults)
* Ward of the state
* Unable to read or write English

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy for glucose management | Baseline, Day 3 of CGM, Day 7 of CGM, Day 14 of CGM, Day 60 of study
  Self-efficacy will be adapted from a validated survey of self-efficacy for type II diabetes management (DMSES UK)

SECONDARY OUTCOMES:
Motivation for glucose management | Baseline, Day 3 of CGM, Day 7 of CGM, Day 14 of CGM, Day 60 of study
  Assessed using items from the Treatment Self-Regulation Questionnaire (TSRQ)
Pregnancy-specific stress | Baseline, Day 60 of study participation
  Pregnancy-specific stress will be measured (via questionnaire) using a validated scale that was empirically associated with birth outcomes
Social support | Baseline, Day 3 of CGM, Day 7 of CGM, Day 14 of CGM, Day 30 of group chat participation, Day 60 of study participation
  A social support survey was adapted from the validated Inventory of Socially Supportive Behaviors (ISSB) that assess multiple subtypes of social support (emotional, informational, instrumental/tangible, belonging, appraisal)
Pre-natal care satisfaction | Baseline, Day 60 of study completion
  Prenatal care satisfaction will be assessed using a combination of questions from Raube and colleague's validated questionnaire and the Mother's Autonomy in Decision Making (MADM) scale. The combination of questionnaires is scored as "Excellent, Good, Average, Poor, N/A".

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided